CLINICAL TRIAL: NCT01560858
Title: A Retrospective Observational Study to Describe Treatment Patterns Among Patients With Prostate Cancer Prior to Diagnosis of a Castration-resistant State, in Routine Clinical Practice in Spain.
Brief Title: Treatment Patterns Among Patients With Prostate Cancer Prior to Diagnosis of a Castration-resistant State
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-92-52014-196
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the protocol is to describe treatment patterns among patients with prostate cancer prior to diagnosis of castration-resistant state.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with prostate cancer who had developed a castration resistant state in the last 24 months prior to starting the study
* Patient must give written informed consent before any study related procedure

Exclusion Criteria:

* Patients with medical histories lacking data required to evaluate the study objectives

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 407 (Actual)
Dates: Start 2012-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Prior treatment before progression to advanced or metastatic disease. | Baseline
  Number of participants with each category of treatment.
Treatment of advanced or metastatic disease. | Baseline
  Number of participants with each category of treatment.

SECONDARY OUTCOMES:
Clinical management of Castration-Resistant Prostate Cancer (CRPC) patients in the clinical practice. | Baseline
  Percentage of specialists (urologist, radiotherapist, oncologist or other specialist) in charge of treatment decision in CRPC patients.
Number of CRPC patients with signs and symptoms of metastatic disease. | Baseline
Time to castration resistant state after beginning of hormonotherapy. | Baseline
Demographic data. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Private practice, La Cañada, Paterna, Valencia, Spain